CLINICAL TRIAL: NCT06990087
Title: CurePML - Allogeneic HPyV-2-specific T-cell Therapy in Patients With Progressive Multifocal Leukoencephalopathy
Brief Title: T-cell Therapy in Patients With PML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CurePML; 01EN2302 (Other Grant/Funding Number: BMBF)
Record Dates: First submitted 2025-04-29; First posted 2025-05-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Progressive Multifocal Leucoencephalopathy (PML)
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Study participants receive complete or partially HLA-matched, allogeneic HPyV-2-specific T-lymphocytes
  Interventions: Drug: Application of T-lymphocytes

INTERVENTIONS:
Drug: Application of T-lymphocytes — Dosage form: Infusion; Route of administration: Intravenous; Cell dose: 1-2 x 10.000 viable CD3+ T-lymphocytes per kg bodyweight; Application at three timepoints: baseline, after two weeks, after 6 weeks

SUMMARY:
There is no approved standard treatment für progressive multifocal leukoencephalopathy (PML). The sponsor of the study is developing a new treatment. For this reason, the investigational medicinal product (IMP) called 'human allogenic HPyV-2-specific T cells' is to be tested in this study. The sponsor wants to find out whether the IMP is safe, influences the neurological status and improves the quality of the life of patients . It is to be investigated whether the IMP can be used to treat the disease and whether it could have an advantage over the standard therapy in terms of survival rate.

DETAILED DESCRIPTION:
Progressive multifocal leukoencephalopathy (PML) is a severe infection of the central nervous system (CNS) caused by reactivation of human polyoma virus 2 (HPyV-2). HPyV-2 usually produces asymptomatic, lifelong persistent or latent infection in the general population. However, in patients with long lasting and profound impairment of cellular immunity, HPyV-2 can reactivate from latency leading to lytic infection of CNS glial cells and thus to encephalitis PML. PML is usually fatal or at least associated with severe disability which makes it a relevant target for the search of appropriate therapeutic options.

The investigational medicinal products (IMPs) under test are fresh and cryopreserved allogeneic HPyV-2-specific T-lymphocyte apheresis concentrates.

Each patient will receive one HPyV-2-specific T-lymphocyte fresh product and two additional cryopreserved products from the same manufacture with the same dose 2 and 6 weeks after baseline, respectively.

This is the first controlled clinical trial to treat patients suffering from PML with this specific methodology of T-cell therapy. The currently available evidence of safety and efficacy is only based on a small series of individual cases treated on a compassionate use basis. This study aims to generate data on safety and first evidence of efficacy within a standardized clinical trial protocol complying to ICH-GCP principles.

ELIGIBILITY:
Inclusion Criteria:

* Adults* aged ≥ 18 years with PML (diagnosed ≤ 60 days before screening) associated with one or more of the following risk factors: lymphoproliferative diseases, immunosuppressive therapy, or lymphopenia
* Signed written informed consent from subject and/or legal representative
* HPyV-2 detection in CSF by PCR analysis or in brain biopsy

Exclusion Criteria:

* PML caused by HIV
* PML caused by natalizumab
* PML occurring within five 5 years after hematopoietic stem-cell transplantation or CAR T cell therapy, or resulting from chronic lymphocytic leukemia (CLL)
* Patients who are unable to follow the study protocol, either on their own or with the support of a reliable representative, will be excluded
* Pregnancy or breastfeeding
* Currently receiving chemotherapy
* Present (within 2 weeks before screening visit) and continuous treatment with immune checkpoint inhibition therapy
* Severe infections other than PML (e.g. sepsis, pneumonia)
* Hypersensitivity to any of the components of the medications used
* Inability to undergo MRI examination (e.g. implanted incompatible medical devices, claustrophobia)
* Participation in another clinical trial (other investigational drugs or devices at the time of enrolment or within 30 days prior to enrolment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Demonstrate efficacy of treatment | 6 months after diagnosis
  Determine proportion of patients surviving 6 months (overall survival) since diagnosis.

SECONDARY OUTCOMES:
Safety assessment | During 12 months from baseline
  Recording of AEs, SAEs, AE of special interest (GvHD, allergic reactions).
Safety assessment | At 12 months from baseline
  Determine proportion of patients surviving 12 months (via telephone interview).
Assessment of potential inflammatory safety concerns | During 6 months from baseline
  Laboratory examination of differential blood count (cells/microliter).
Assessment of potential inflammatory safety concerns | During 6 months from baseline
  Laboratory examination of c-reactive protein (CRP; mg/l).
Assessment of potential inflammatory safety concerns | During 6 months from baseline
  Laboratory examination of serum-immunoglobulin G (IgG; g/l).
Safety assessment of potential electrolyte imbalance | During 6 months from baseline
  Laboratory examination of potassium, sodium (mmol/l).
Safety assessment of potential renal dysfunction | During 6 months from baseline
  Laboratory examination of creatinine (micromol/l).
Safety assessment of potential renal dysfunction | During 6 months from baseline
  Laboratory examination of urea (mmol/l).
Safety assessment of potential liver dysfunction | During 6 months from baseline
  Laboratory examination of aspartate aminotransferase (AST; U/l), alanine aminotransferase (ALT; U/l).
Safety assessment of potential liver dysfunction | During 6 months from baseline
  Laboratory examination of bilirubin (micromol/l).
Safety assessment of potential coagulation disorder | During 6 months from baseline
  Laboratory examination of coagulation parameters (prothrombin time (INR; ratio).
Safety assessment of potential coagulation disorder | During 6 months from baseline
  Laboratory examination of partial thromboplastin time (PTT; sec.).
Rate of development of IRIS | During 6 months from baseline
  Evaluate possible development of immune reconstitution inflammatory syndrome (IRIS) by MRI of the brain and clinical examination.
Assessment of neurological status by Modified Rankin Scale (mRS) | Change from baseline after 6 months
  mRS compromising 6 levels of degree of impairment (minimum 0 = no symptoms, maximum 6 = death).
Assessment of neurological status by Karnofsky Performance Status Index | Change from baseline after 6 months
  Karnofsky Performance Status Index compromising 11 levels of functional impairment (minimum 100% = no symptoms, maximum 0% = death).
Assessment of neurological status by Montreal Cognitive Assessment (MoCA) | Change from baseline after 6 months
  Montreal Cognitive Assessment (MoCA) compromising 8 categories to detect cognitive impairment (minimum 0 points, maximum 30).
Determine change in viral load | Change from baseline after 6 months
  HPyV-2 viral load in CSF quantified by PCR.
Evaluation of quality of life improvements by quality of life questionnaire (EQ-5D-5L) | Change from baseline after 6 months
  Quality of life questionnaire (EQ-5D-5L) compromising 5 categories to determine quality of life (minimum 0%, maximum 100%).
Analysis of immunological response | Change from baseline after 6 months
  HPyV-2specific -T-lymphocyte frequency in blood detected by IFN-gamma cytokine secretion.
Determine lesion volume | Change from baseline after 6 months
  Determine lesion volume on brain MRI.
Evaluation of survival | At month 12
  Evaluation of survival by telephone interview.

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - LMU Klinikum Campus Großhadern, München, Bavaria
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Hannover Medical School, Hanover, Lower Saxony
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein